CLINICAL TRIAL: NCT07077434
Title: A Phase 1 Open-Label, Multi-Center Study to Evaluate Pharmacokinetics, Safety and Tolerability of BMS-986504 in Japanese and Chinese Participants With Advanced Solid Tumors With Homozygous MTAP Deletion
Brief Title: A Study to Assess Safety, Tolerability and Drug Levels of BMS-986504 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA240-0010
Record Dates: First submitted 2025-07-21; First posted 2025-07-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: MTAP; PRMT5; MRTX1719; CDKN2A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMS-986504 Arm (Experimental)
  Interventions: Drug: BMS-986504

INTERVENTIONS:
Drug: BMS-986504 — Specified dose on specified days
  Other Names: MRTX1719

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and drug levels of BMS-986504 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of a solid tumor malignancy with homozygous deletion of the MTAP gene detected in tumor tissue.
* Participants must have unresectable or metastatic disease not amenable to curative therapies after progression on prior therapies at the time of enrollment.
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must have presence of at least one measurable tumor lesion per RECIST 1.1 at baseline.

Exclusion Criteria:

* Participants must not have prior treatment with a Protein arginine methyltransferase 5 (PRMT5) or Methionine adenosyltransferase 2A (MAT2A) inhibitor.
* Participants must not have active brain metastases or carcinomatous meningitis.
* Participants must not have a history of gastrointestinal disease or other gastrointestinal conditions (e.g., uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications.
* Participants must not have known severe hypersensitivity to study treatment and/or any of its excipients.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-01-19 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of BMS-986504 | Up to approximately Day 64
Time to Reach Maximum Plasma Concentration (Tmax) of BMS-986504 | Up to approximately Day 64
Area Under Curve (AUC) of BMS-986504 | Up to approximately Day 64
Mean Elimination Half-life (T-HALF) of BMS-986504 | Up to approximately Day 64
Apparent Total Body Clearance (CLT/F) of BMS-986504 | Up to approximately Day 64
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of BMS-986504 | Up to approximately Day 64

SECONDARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) | Up to approximately Day 25
Number of Participants With Treatment-related Adverse Events (AE) | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With all-cause AEs | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With Treatment-related Serious AEs (SAEs) | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With all-cause SAEs | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With AEs Leading to Dose Interruption | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With AEs Leading to Dose Reduction | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With AEs Leading to Treatment Discontinuation | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With AEs Leading to Death | Up to approximately 28 days after last dose of BMS-986504
Number of Participants With Laboratory Abnormalities | Up to approximately 28 days after last dose of BMS-986504

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- China (8):
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Local Institution - 0006, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
- Japan (4):
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html